CLINICAL TRIAL: NCT03012841
Title: STOP Persistent AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOP Persistent AF
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Arctic Front Advance Cardiac CryoAblation Catheter and Freezor MAX Cardiac CryoAblation Catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects enrolled and treated with Arctic Front Advance Cardiac CryoAblation Catheter
  Interventions: Device: Arctic Front Advance Cardiac CryoAblation Catheter

INTERVENTIONS:
Device: Arctic Front Advance Cardiac CryoAblation Catheter — Cryoablation
  Other Names: Freezor MAX Cardiac CryoAblation Catheter

SUMMARY:
To demonstrate safety and effectiveness of the Arctic Front Advance™ and Freezor MAX® Cardiac CryoAblation Catheters for the treatment of drug refractory recurrent symptomatic persistent atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Documentation of symptomatic persistent AF: Defined as having a continuous episode lasting longer than 7 days but less than 6 months documented by consecutive ECG recordings OR Defined as having a continuous episode lasting longer than 7 days but less than 6 months documented by an ECG recording and one doctor note indicating patient had symptoms consistent with AF
* Failure or intolerance of at least one Class I or III antiarrhythmic drug
* Age 18 or older (or older than 18 if required by local law)

Exclusion Criteria:

* Left atrial diameter > 5.0 cm (anteroposterior)
* Prior left atrial ablation or surgical procedure (including left atrial appendage closures)
* Presence or likely implant of a permanent pacemaker, biventricular pacemaker, loop recorder, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) within 12 months
* Presence of any pulmonary vein stents
* Presence of any pre-existing pulmonary vein stenosis
* Pre-existing hemidiaphragmatic paralysis
* Presence of any cardiac valve prosthesis
* +3 and +4 mitral valve regurgitation or stenosis
* Any cardiac surgery, myocardial infarction, percutaneous coronary intervention (PCI) / percutaneous transluminal coronary angioplasty (PTCA) or coronary artery stenting which occurred during the 3 month interval preceding the consent date
* Unstable angina
* New York Heart Association (NYHA) Class III or IV congestive heart failure and/or documented left ventricular ejection fraction (LVEF) less than or equal to 35% measure by acceptable cardiac testing (e.g. Transthoracic echocardiogram (TTE))
* Primary pulmonary hypertension
* Rheumatic heart disease
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* Active systemic infection
* Hypertrophic cardiomyopathy
* Cryoglobulinemia
* Uncontrolled hyperthyroidism
* Any cerebral ischemic event (strokes or transient ischemic attacks (TIAs)) which occurred during the 6 month interval preceding the consent date
* Any woman known to be pregnant or breastfeeding, or any woman of child bearing potential who is not on a reliable form of birth regulation method or abstinence
* Life expectancy less than one year
* Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of the study not pre-approved by Medtronic
* Known allergies or hypersensitivities to adhesives
* Known drug or alcohol dependency
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Calkins, MD, Principal Investigator — Johns Hopkins University; Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (25):
- United States (19):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Cardiac Arrhythmia Service, Boca Raton, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Luke's Health System, Kansas City, Missouri
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Northwell Health (Lenox Hill Hospital and Staten Island University Hospital), New York, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Canada (3):
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec
- Japan (3):
  - Tokyo Medical and Dental University, Bunkyō, Tokyo
  - Jikei University Hospital, Tokyo
  - Yokohama City Minato Red Cross Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su WW, Reddy VY, Bhasin K, Champagne J, Sangrigoli RM, Braegelmann KM, Kueffer FJ, Novak P, Gupta SK, Yamane T, Calkins H; STOP Persistent AF Investigators. Cryoballoon ablation of pulmonary veins for persistent atrial fibrillation: Results from the multicenter STOP Persistent AF trial. Heart Rhythm. 2020 Nov;17(11):1841-1847. doi: 10.1016/j.hrthm.2020.06.020. Epub 2020 Jun 24. PMID 32590151

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified Intent to Treat (mITT) Group: Subjects enrolled and treated with Arctic Front Advance Cardiac CryoAblation Catheter
- Not Treated: Subjects enrolled, but not treated with an Arctic Front Advance Cryoablation catheter.
Period: Overall Study
Arm/Group | Modified Intent to Treat (mITT) Group | Not Treated
Started | 165 | 21
Completed | 145 | 0
Not Completed | 20 | 21
Not completed — Protocol Violation | 0 | 10
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Unable to complete 12 month visit | 6 | 0
Not completed — Subject relocation | 1 | 0
Not completed — Seasonal winter travel | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — No ablation performed | 0 | 2
Not completed — Study reached n=165 treated subject cap | 0 | 5
Not completed — Insurance change | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes those subjects who were enrolled and underwent ablation with an Arctic Front Advance CryoAblation catheter.
Groups:
- Modified Intent to Treat Group (mITT): Subjects enrolled and treated with Arctic Front Advance Cardiac CryoAblation Catheter
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 116
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 142
  Japanese | 15
  Black | 2
  Filipino | 1
  Other Asian | 1
  Subject/physician chose not to provide | 4
Region of Enrollment [Number; unit: participants]
  Canada | 30
  United States | 120
  Japan | 15
Time from Persistent Atrial Fibrillation (AF) Onset [Mean (Standard Deviation); unit: years] | 0.6 (1.4)
Duration of Longest Persistent AF Episode [Median (Full Range); unit: days] | 60.9 [7 to 182.6]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Free From Treatment Failure at 12 Months After the Pulmonary Vein Isolation (PVI) Ablation Procedure.
Description: Treatment failure is defined as any of the following components:
  * Acute procedural failure
  * Documented AF/atrial tachycardia (AT)/atrial flutter (AFL) after the 90 day blanking period
  * A reablation for the treatment of recurrent AF/AT/AFL after the 90 day blanking period
  * Class I or III antiarrhythmic drug (AAD) dose increase from the historic maximum ineffective dose (prior to the ablation procedure) or initiation of a new Class I or III AAD after the 90 day blanking period.
  * Ablation using radiofrequency (RF) in the left atrium
  Blanking period is defined as the first 90 days after the index ablation procedure.
  Acute procedural failure is defined as:
  * Inability to isolate all accessible targeted pulmonary veins (minimally assessed for entrance block and, where assessable, exit block) during the index procedure
  * Left atrial non-PVI ablations including but not limited to, ablation of linear lesions complex fractionated electrograms or non-PV triggers
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 165
percentage of participants | 54.8 [46.7 to 62.1]
Statistical Analysis 1: Comparison: Modified Intent to Treat Group (mITT); Test type: Superiority — The formal alternative hypothesis test for the primary effectiveness objective was that the Kaplan-Meier estimator of treatment success at 12 months (365 days) was greater than 40%, against the null hypothesis that it was less than or equal to 40%; p < 0.001, Exact binomial; Exact binomial p-value is shown, but the confidence intervals reported are calculated from Greenwood's approximation of the standard error; Kaplan-Meier (product-limit) estimator = 54.8, 95% CI 2-sided [46.7 to 62.1]

2. Primary Outcome: Percent of Subjects Free From a Primary Safety Event at 12 Months After the Pulmonary Vein Isolation (PVI) Ablation Procedure.
Description: A primary safety event is defined as a serious procedure-related or serious system-related adverse event including the following:
  * Transient ischemic attack (within 7 days of ablation procedure)
  * Cerebrovascular accident (within 7 days of ablation procedure)
  * Major bleeding that requires transfusion (within 7 days of ablation procedure)
  * Cardiac perforation, tamponade or pericardial effusion (within 7 days of ablation procedure)
  * Pulmonary vein stenosis (> 75% reduction within 12-months of ablation procedure)
  * Myocardial infarction (within 7 days of ablation procedure)
  * Phrenic nerve injury (unresolved at 12-months)
  * Atrio-esophageal fistula (within 12-months of ablation procedure)
  * Death (within 7 days of ablation procedure)
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 165
percentage of participants | 0.6 [0.1 to 4.4]
Statistical Analysis 1: Comparison: Modified Intent to Treat Group (mITT); Test type: Superiority — The formal alternative hypothesis tested for the primary safety objective was that the Kaplan-Meier estimator of the proportion of subjects with primary safety events at 12 months (365 days) was less than 13%, against the null hypothesis that it was greater than or equal to 13%; p = 0.002, Exact binomial; [statistical method as in outcome 1, analysis 1]; Kaplan-Meier (product-limit) estimator = 0.6, 95% CI 2-sided [0.1 to 4.4]

3. Secondary Outcome: Change in Quality of Life Between Baseline and 12 Months: Atrial Fibrillation Effect on QualiTy-of-life (AFEQT)
Description: Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire completed at baseline and 12 month visits. The AFEQT instrument yields scores from 0 (representing the worst possible debilitation from AF) to 100 (representing no reduction in quality of life from AF).
Time Frame: Baseline and 12 months
Population: Treated subjects completing at least 50% of questions on AFEQT questionnaires at both baseline and 12-month visits
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Treated 12-month Completers: Subjects enrolled and treated with Arctic Front Advance Cardiac CryoAblation Catheter who had complete QoL questionnaires at baseline and follow-up
Arm/Group | Treated 12-month Completers
Number analyzed (Participants) | 141
score on a scale | 25.8 [22.1 to 29.5]
Statistical Analysis 1: Comparison: Treated 12-month Completers; The formal alternative hypothesis tested was that the mean 12-month change in AFEQT composite scores was greater than 0, against the null the hypothesis that it was equal to 0; Test type: Superiority; p < 0.001, t-test, 1 sided — A Hommel multiple testing procedure was utilized to maintain overall alpha of 0.025 for the 3 hypotheses tested for the secondary objective; Mean Difference (Net) = 25.8, 95% CI 2-sided [22.1 to 29.5]

4. Secondary Outcome: Change in Quality of Life Between Baseline and 12 Months: Medical Outcome Study Short Form-12 (SF-12) Physical Component
Description: Medical Outcome Study Short Form-12 (SF-12) questionnaire completed at baseline and 12 month visits. The SF-12 instrument has two composite scores, one for physical health and one for mental health. Each yields scores from 0 (representing the worst possible debilitation) to 100 (representing no reduction in quality of life).
Time Frame: Baseline and 12 months
Population: Treated subjects fully completing SF-12 questionnaires at both baseline and 12-month visits
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treated 12-month Completers
Number analyzed (Participants) | 142
score on a scale | 5.0 [3.5 to 6.5]
Statistical Analysis 1: Comparison: Treated 12-month Completers; The formal alternative hypothesis tested was that the mean 12-month change in SF-12 physical composite scores was greater than 0, against the null the hypothesis that it was equal to 0; Test type: Superiority; p < 0.001, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 5.0, 95% CI 2-sided [3.5 to 6.5]

5. Secondary Outcome: Change in Quality of Life Between Baseline and 12 Months: Medical Outcome Study Short Form-12 (SF-12) Mental Component
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: Treated subjects fully completing SF-12 questionnaires at both baseline and 12-month visits
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treated 12-month Completers
Number analyzed (Participants) | 142
score on a scale | 4.9 [3.2 to 6.6]
Statistical Analysis 1: Comparison: Treated 12-month Completers; The formal alternative hypothesis tested was that the mean 12-month change in SF-12 mental composite scores was greater than 0, against the null the hypothesis that it was equal to 0; Test type: Superiority; p < 0.001, t-test, 1 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 4.9, 95% CI 2-sided [3.2 to 6.6]

ADVERSE EVENTS:
Time Frame: All adverse events were collected between subject consent (enrollment) and study completion (1 year post study cryoablation procedure)
Groups:
- Enrolled Subjects: All enrolled and consented subjects
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/186
Serious Adverse Events (participants affected / at risk) | 34/186
Other Adverse Events (participants affected / at risk) | 52/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=186)
Atrial fibrillation (Cardiac disorders) | 10 (11)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic perforation (Vascular disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Puncture site haematoma (General disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=186)
Atrial fibrillation (Cardiac disorders) | 44 (62)
Atrial flutter (Cardiac disorders) | 20 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principle Investigator (PI) agrees they will not independently discuss or publish trial results until a multi-center publication is released. If a multi-center publication is not released within one year after completion of the Study at all Study sites, PIs will have the right to publish the results of and information pertaining to their activities. Any such Publication must be submitted to Medtronic for review and comment at least sixty (60) days prior to submission or presentation.

DOCUMENTS (4):
  • Study Protocol: Version 4 (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03012841/Prot_001.pdf
  • Study Protocol: Version 5 (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03012841/Prot_002.pdf
  • Study Protocol: Version 6 (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT03012841/Prot_003.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03012841/SAP_000.pdf